CLINICAL TRIAL: NCT00884013
Title: Program Evaluation of New York City Health eHearts Pay for Quality Program
Brief Title: New York City (NYC) Health eHearts Pay for Quality Pilot
Acronym: ehearts
Status: Completed | Type: Observational
Sponsor: New York City Department of Health and Mental Hygiene (Other Government)
Collaborators: Robin Hood Foundation (Unknown)
Responsible Party: Farzad Mostashari/Assistant Commission, NYC DOHMH
Other Study IDs: PCIP001
Record Dates: First submitted 2009-04-16; First posted 2009-04-20 (Estimated); Last update posted 2009-04-20 (Estimated); Status verified 2009-04

CONDITIONS: Hypertension; Diabetes; Smoking; Ischemic Cardiovascular Disease
Keywords: Pay for Quality; Provider; Clinical Decision Support; Quality Reporting; Quality Measurement
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- 1: Quality Payment and all clinical reminders turned on
- 2: Quality Payment and ABCS measures reminders turned on
- 3: Quality Payment and non-ABCS measures reminders turned on
- 4: Quality Reporting and Recognition with all clinical reminders turned on
- 5: Quality Reporting and Recognition with ABCS measures reminders turned on
- 6: Quality Reporting and Recognition with non-ABCS measures reminders turned on

SUMMARY:
Do monetary incentives in small independent primary care practices improve the delivery of preventive services as recommended by U.S. Preventive Services Task Force (USPSTF) guidelines for cardiovascular health?

DETAILED DESCRIPTION:
The NYC DOHMH received a private donation from the Robin Hood Foundation to provide monetary incentives to small practices for improving their delivery of preventive services in neighborhoods experiencing health disparities.

Practices recruited by NYC DOHMH to adopt an electronic health record will be randomized to receive monetary incentives for improving both patient outcomes and delivery of care on: aspirin therapy, blood pressure control, cholesterol control, and smoking cessation intervention. The set of quality measures are referred to the ABCS.

The NYC DOHMH will be collecting provider surveys on their experience on quality measurement and participation in other pay-for-performance programs, as well as transmit aggregated information on their performance on the ABCS to DOHMH on a monthly basis.

ELIGIBILITY:
Inclusion Criteria:

* Primary Care Providers

Exclusion Criteria:

* Specialists
* Pediatricians
* Obstetricians
* Gynecologists

Min Age: 22 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Adult Primary Care Providers that have adopted an electronic health record in New York City in non-hospital based practices.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2009-01

PRIMARY OUTCOMES:
percent of patients eligible for quality measures (ABCS) | 1 year

SECONDARY OUTCOMES:
use of EHR clinical reminders | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Farzad Mostashari, MD, MPH, Principal Investigator — NYC DOHMH
Locations (1):
- New York City Departemnt of Health and Mental Hygiene, New York, New York, United States

REFERENCES:
- [Derived] Bardach NS, Wang JJ, De Leon SF, Shih SC, Boscardin WJ, Goldman LE, Dudley RA. Effect of pay-for-performance incentives on quality of care in small practices with electronic health records: a randomized trial. JAMA. 2013 Sep 11;310(10):1051-9. doi: 10.1001/jama.2013.277353. PMID 24026600